CLINICAL TRIAL: NCT02919449
Title: Phase 1 Dose Escalation Trial of Intra-Tumoral Injection of Sodium Iodide Simporter (NIS) Measles Virus (Edmonston Strain) in Combination With Atezolizumab in Patients With Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Dose Escalation Trial of Intra-Tumoral Injection of NIS Measles Virus in Combination With Atezolizumab
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Vyriad, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VYR-MV1-101
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2022-01

CONDITIONS: Recurrent Non-Small Cell Lung Cancer
Keywords: Lung Cancer Measles Nivolumab Opdivo
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MV-NIS and Atezolizumab (Experimental): MV-NIS will be administered intratumorally as a single dose on day 1. Atezolizumab will be given at day 15 and then every 3 weeks.
  Interventions: Biological: MV-NIS; Biological: Atezolizumab

INTERVENTIONS:
Biological: MV-NIS — This is an open label single ascending dose phase I study designed to determine the safety profile and MTD after IT administration of a single dose of MV-NIS in combination with Atezolizumab in patients with metastatic NSCLC
Biological: Atezolizumab — Atezolizumab will be administered every 3 weeks

SUMMARY:
This a Phase 1 study designed to determine the maximum tolerated dose (MTD) and toxicity of attenuated Measles virus (MV-NIS) combined with Atezolizumab in patients with recurrent and metastatic NSCLC.

DETAILED DESCRIPTION:
Phase 1, dose escalation study of the combination of intra-tumoral MV-NIS and systemic atezolizumab in patients with recurrent and metastatic NSCLC. After the dose escalation phase of the trial, a dose expansion cohort was planned to further investigate safety, clinical and immune responses at the MTD. A standard 3+3 design was to be used for the dose escalation part of the study. Starting at dose level 1, three patients were to be treated per dose level. MV-NIS was to be administered once intra-tumorally (IT) on Day 1 of treatment in 3 escalating dose cohorts, starting at dose level 1 x 10e8

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of metastatic lung cancer, with histologic confirmation of the primary NSCLC histology and with at least one lesion amenable for intra-tumoral injection of MV-NIS.
* Patient meets the FDA-approved indication for Atezolizumab treatment in NSCLC.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
* Ability to provide informed consent.
* Adequate hematological, liver and kidney function.
* Must be willing to implement contraception throughout study and for the 8 weeks following last study drug administration.

Key Exclusion Criteria:

* Any of the following prior therapy: Chemotherapy ≤ 3 weeks prior to registration. Biologic therapy ≤ 4 weeks prior to registration. Radiation therapy ≤ 3 weeks prior to registration
* Other concurrent investigational therapy (utilized for a non-FDA-approved indication and in the context of a research investigation).
* Pregnant women.
* Nursing women.
* Men or women of childbearing potential who are unwilling to employ adequate contraception during treatment and 8 weeks following the completion of study drug treatment.
* Allergy to measles vaccine or history of severe reaction to prior measles vaccination.
* History of organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Bexon, MD, Study Director — Vyriad, Inc.
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MV-NIS and Atezolizumab: MV-NIS will be administered intratumorally as a single dose on day 1. Atezolizumab 1200 mg IV will be given at day 15 and then every 3 weeks.
  MV-NIS: This is an open label single ascending dose phase I study designed to determine the safety profile and MTD after IT administration of a single dose of MV-NIS in combination with Atezolizumab in patients with metastatic NSCLC
  Atezolizumab: Atezolizumab will be administered every 3 weeks
Period: Overall Study
Arm/Group | MV-NIS and Atezolizumab
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Investigator decision | 1

BASELINE CHARACTERISTICS:
Population: A maximum of 21 patients were planned for this study, 2 patients were treated prior to the closure of the study. The study was closed for administrative reasons.
Arm/Group | MV-NIS and Atezolizumab
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of MV-NIS in Combination With Atezolizumab
Description: To determine the maximum tolerated dose (MTD) of the intra-tumoral administration of an Edmonston strain MV genetically engineered to produce NIS (MV-NIS), in combination with the PD-L1 inhibitor atezolizumab
Time Frame: 28 days after MV-NIS administration for each dose cohort
Population: The study was prematurely closed for administrative reasons. The very limited number of patients (n=2) and short duration of study treatment does not allow any meaningful conclusions to be drawn from the available data.
Arm/Group | MV-NIS and Atezolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AE data was collected from when the patient was enrolled in the study starting from the day of informed consent until 30 days after the last dose of study drug or the patient withdraws from the study. Event reporting occurred over a total period of 3 months (23August 2017-09Nov2017), the duration of the study.
Arm/Group | MV-NIS and Atezolizumab
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MV-NIS and Atezolizumab (N=2)
Chills (Infections and infestations) | 2 (2)
Viral illness (Infections and infestations) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausa (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was closed prematurely due to administrative reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-03): https://cdn.clinicaltrials.gov/large-docs/49/NCT02919449/Prot_SAP_000.pdf